CLINICAL TRIAL: NCT05795894
Title: Suicidology and Anthropology Research Protocol : Qualitative Study of Suicidal Recrudescence Among Adolescents in November 2021
Brief Title: Qualitative Study of Suicidal Recrudescence Among Adolescents in November 2021
Acronym: Suicide-Covid
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondation Lenval (Other)
Responsible Party: Sponsor
Other Study IDs: 22-HPNCL-07
Record Dates: First submitted 2023-03-21; First posted 2023-04-03 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Suicide; COVID-19
Keywords: pediatric
MeSH Terms: conditions — Suicide; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patents: Questionnaires
  Interventions: Behavioral: STAI-Y; Behavioral: BDI scale; Behavioral: M.I.N.I.Kid; Behavioral: PCL-5

INTERVENTIONS:
Behavioral: STAI-Y — Situational Anxiety and Trait Anxiety Inventory
Behavioral: BDI scale — • Beck Depression Inventory scale
Behavioral: M.I.N.I.Kid — Suicidal risk" module of the Mini-International Neuropsychiatric Interview child/adolescent version
Behavioral: PCL-5 — Post-traumatic Check List Scale

SUMMARY:
A qualitative study, combining psychiatric and anthropological perspectives, focused on the lived experiences of patients who had recourse to HPNCL emergencies during the period of November 2021, as well as the experiences and perceptions of those around them - such as their family, teachers or school and nursing staff. This multi-site approach will provide a multidimensional perspective on the experience of individuals and those around them, as well as a triangulation of data.

The hypotheses to explain the increase in the rate of suicidal crisis will be addressed through semi-structured interviews proposed to the participants of the study.

DETAILED DESCRIPTION:
Interviews in the presence of two members of the research team (child psychiatrists, psychologists, anthropologists, etc.) will be offered to participants. These interviews will be face-to-face when possible, but can also be done remotely, by teleconsultation, depending on the preferences of the participants.

These interviews will be based on a questionnaire established beforehand evoking the history of mental disorders and the experience of the participant in the study and his entourage of the Covid-19 health crisis.

All information exchanged during these interviews will be made anonymous (data collected and processed as well as the results presented). They will be used exclusively in the context of the study and not communicated to the medical team involved in the patient's care.

The proposed interviews will be carried out separately with:

* The patient who consulted the emergency room during the month of November 2021
* The parent(s) of the study participant
* One or more health professionals taking care of the patient
* The school attended by the patient who will be questioned about the suicidal problem and Covid-19 in general or not about the patient in particular.
* Child welfare professionals (ASE) potentially involved in the care of the study participant.

Questionnaires will also be carried out with patients in order to complete the assessment of their clinical condition at a distance from the psychological crisis:

ELIGIBILITY:
Inclusion Criteria:

* Any patient having consulted in the child psychiatric emergency room of the HPNCL between November 1, 2021 and November 30, 2021 for suicidal thoughts.
* Age between 13 years and 17 years and 11 months
* Good understanding of written and oral French
* Collection of the informed consent of the patient and of one of the two parents or holder of parental authority

Exclusion Criteria:

* Inability to comply with the instructions defined and exposed during inclusion
* Refusal of participation by the patient or one of the legal guardians

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: * The patient who consulted the emergency room during the month of November 2021
  * The parent(s) of the study participant
  * One or more health professionals taking care of the patient
  * The school attended by the patient who will be questioned about the suicidal problem and Covid-19 in general or not about the patient in particular.
  * Child welfare professionals (ASE) potentially involved in the care of the study participant
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2022-07-12 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Situational Anxiety and Trait Anxiety Inventory | at inclusion
  This inventory aims to assess anxiety as a "personality trait" (feelings of apprehension, tension, nervousness and worry that the subject usually feels), and anxiety as a ' "emotional state" linked to a particular situation (feelings of apprehension, tension or nervousness that the subject feels at a specific moment).
  This is a questionnaire comprising 20 items for the "state" form and 20 items for the "trait" form. The instruction is to answer "in general, in the usual way" for the "trait" scale and "at the moment" for the "state" scale.
  Each score can therefore vary from 20 to 80 with a "very high" anxiety norm when the threshold is > 65, "high" between 56 and 65, "medium" between 46 and 55, "low" between 36 and 45 and "very low" for a score < or = 35.

SECONDARY OUTCOMES:
Beck Depression Inventory | at inclusion
  The Beck Depression Inventory is a diagnostic self-questionnaire allowing a quantitative estimation of the intensity of depressive symptoms in adults and adolescents. It consists of 21 symptom and attitude items, which describe a specific behavioral manifestation of depression, graded from zero to three by a series of four statements reflecting the degree of severity of the symptom. The subject must indicate, among the propositions, the one that best describes how he has felt during the last seven days. The total score varies between 0 (absence of depressive symptoms) and 63. Some authors suggest that in a normal population, a total BDI score greater than 15 is an argument in favor of depression. The results of this scale can also be categorized according to: normal score < 15; mild depression: 10 to 18; moderate depression: 19 to 29; severe depression > 30
"Suicidal risk" module of the Mini-International Neuropsychiatric Interview child/adolescent | at inclusion
  The MINI is a short structured diagnostic interview, jointly developed by psychiatrists and clinicians in the United States and Europe, for DSM IV and CIM 10 psychiatric disorders. It was designed to meet the need for a short structured psychiatric interview for clinical trials and epidemiological studies and for use as a first step in monitoring outcomes in clinical settings. Its very brief "suicide risk" module is sometimes used alone to determine the level of suicide risk. It is composed of 6 binary questions. The level of risk is established according to the number of questions having obtained a positive answer
Post-traumatic Check List Scale | at inclusion
  The questionnaire includes 20 items, each question is to be rated between 1 and 5 depending on the intensity and frequency of symptoms during the previous month. The maximum score is 80. A threshold of 33 to 38 is proposed for screening for post-traumatic stress disorder (PTSD)

CONTACTS AND LOCATIONS:
Overall Officials: Louise-Emilie DUMAS, MD, Principal Investigator — Fondation Lenval
Locations (1):
- hôpital Lenval, Nice, France